CLINICAL TRIAL: NCT00627510
Title: Routine Plasma Level Determination to Compare Actual vs Expected Plasma Levels at Psychiatric Inpatient Admission for Determination of Compliance and/or Speed of Drug Metabolism
Brief Title: Routine Plasma Level Determination to Compare Actual vs Expected Plasma Levels at Psychiatric Inpatient Admission
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Gerald Zernig, Assoc.Prof.Pharmacology, Medical University Innsbruck
Other Study IDs: PMUPSY20050001
Record Dates: First submitted 2008-02-22; First posted 2008-03-03 (Estimated); Last update posted 2008-03-03 (Estimated); Status verified 2008-02

CONDITIONS: Depression; Affective Disorders, Psychotic
Keywords: Therapeutic Drug Monitoring (TDM); Antidepressant; Antipsychotic; Treatment adherence; Compliance; Metabolism; Do patients take their psychiatric medication as prescribed?; Do psychiatric patients metabolize their medication faster than expected?; What are the exact odds that the patient of a physician prescribing antidepressants or antipsychotics has plasma levels that are BELOW those intended?
MeSH Terms: conditions — Depression; Affective Disorders, Psychotic; Treatment Adherence and Compliance; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: all patients consecutively admitted to psychiatric inpatient treatment (naturalistic sample from routine psychiatric hospital intake)
  Interventions: Other: Routine psychiatric inpatient treatment

INTERVENTIONS:
Other: Routine psychiatric inpatient treatment — Routine psychiatric inpatient treatment. This is not an interventional study.

SUMMARY:
Compliance with treatment is notoriously low in psychiatric patients. Traditional methods of monitoring compliance, however, may underreport nonadherence to treatment. In this study, actual plasma levels at admission - which are ROUTINELY taken at the Dept Psychiatry of the Paracelsus Medical University - were compared to plasma levels that can be expected from the prescribed preadmission dosing regimen. This was done to give treating psychiatrists a quantitatively precise idea of how frequently they can expect their patients to have plasma levels that are below the level of medication as intended by the prescribing physician.

DETAILED DESCRIPTION:
Context Noncompliance or incomplete compliance with psychopharmacological medication by psychiatric patients is a frequent risk and may be underreported by classical methods (e.g., pill counts or coloring additives).

Objective To determined the prevalence of incomplete compliance and/or faster-than average elimination of the medication by comparing actual plasma levels with those expected from the prescribed dosage under naturalistic routine conditions.

Design Forty-five day prospective routine survey.

Setting University acute inpatient clinic.

Participants All consecutive admissions for acute inpatient treatment from June 1, 2005 to July 15, 2005 who had been treated with antidepressants and/or antipsychotics.

Intervention Determination of plasma levels of all psychiatric medications and their comparison to the expected plasma levels, based on known preadmission dosing regimen and average pharmacokinetic data.

Main outcome measures The percentage of admissions with actual plasma level that were (a) more than 2-fold lower or (b) more than 2-fold higher than the expected plasma level or (c) differing only 0.5- to 2-fold from the expected plasma level.

ELIGIBILITY:
Inclusion Criteria:

* eligible for psychiatric inpatient treatment

Exclusion Criteria:

* not eligible for psychiatric inpatient treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients consecutively admitted for routine psychiatric inpatient treatment
Sampling Method: Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2005-06; Primary Completion 2005-07 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The percentage of admissions with actual plasma level that were (a) more than 2-fold lower or (b) more than 2-fold higher than the expected plasma level or (c) differing only 0.5- to 2-fold from the expected plasma level. | at admission to psychiatric inpatient treatment

SECONDARY OUTCOMES:
There is NO secondary outcome measure. | at admission

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Zernig, MD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Department of Psychiatry I, Paracelsus Medical University, Salzburg, Salzburg, Austria